CLINICAL TRIAL: NCT04556188
Title: The Clinical Influence of Developing a Sustainable Cardiac Surgery Service to Reduce the Burden of Rheumatic Heart Disease in Sub-Saharan Africa
Acronym: RHD-CaSS
Status: Recruiting | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Haukeland University Hospital (Other); Addis Ababa University (Other)
Responsible Party: Sponsor
Other Study IDs: AISCaSS
Record Dates: First submitted 2020-03-17; First posted 2020-09-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Rheumatic Heart Disease; Anticoagulant Adverse Reaction
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: RHD patients undergoing Cardiac surgery at Addis Abeba University Hospital
  Interventions: Procedure: Cardiac surgery
- RHD controls: RHD patients not offered Cardiac surgery
- Anticoagulation controls: Norwegian patients on anticoagulant therapy due to mechanical valve implants

INTERVENTIONS:
Procedure: Cardiac surgery
  Groups: Cases

SUMMARY:
In this bi-directional program of education, training and research activities based on sustainable development goals aim is to develop cardiac surgery service in Ethiopia.

The aim is to evaluate the short and long-term outcome of cardiac surgery for rheumatic heart disease in a low-income country compared to individuals not offered cardiac surgery due to limited availability of the service. Second aim is to evaluate the quality of anticoagulant therapy in patients after cardiac surgery for rheumatic heart disease in a low-income country .

DETAILED DESCRIPTION:
Our objectives are:

1. To evaluate the 30- and 180-days outcome of cardiac surgery for rheumatic heart disease (RHD), and impact of gender, age, clinical findings and echocardiographic classification, during the time of development of cardiac surgery at Black Lion hospital, Ethiopia, in comparison with matched individuals (from the same waiting list) which had no offer of surgery due to limited availability.
2. To evaluate the quality of anticoagulation therapy after cardiac surgery at Black Lion hospital, Ethiopia by evaluating the patients proportion of time in therapeutic INR-level, complications as valve dysfunction, bleeding and thrombosis compared to control patients undergoing valvular replacement due to RHD at Norwegian hospitals.

Population: Approximately 50 RHD patients operated by Our team at Addis Abeba University Hospital, Ethiopia.

Follow up for 180-days for objective 1 and continous follow-up for objective 2. Comparison With matched Controls. Outcome measures: Mortality, complications (heart failure, arrhythmias, thrombosis, bleedings, stroke, infections)

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery due to rheumatic heart disease at the governmental Black Lion University Hospital during the bi-directional programme of education, training and Research to establish Cardiac surgery service

Exclusion Criteria:

* Not willing or able to provide written informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Patients offered Cardiac surgery due to indication symptomatic rheumatic heart disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Short term outcome | 180 days
  Freedom from Death or complication

OTHER OUTCOMES:
Time in therapeutic INR | 2 years
  Time in therapeutic window (anticoagulation)
Mitral valve area by Doppler | 14 days
  Influence of concomitant pathology for Echocardiographic assessment of mitral stenosis
Mitral phenotype in rheumatic heart disease | 0 days
  Influence of mitral valve phenotype with cardiac morphology and complications in untreated rheumatic heart disease patients

CONTACTS AND LOCATIONS:
Locations (4):
- Black Lion University Hospital, Addis Ababa, Ethiopia
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided
No written plan. Under discussion.

REFERENCES:
- [Result] Hauge SW, Dalen H, Estensen ME, Persson RM, Abebe S, Mekonnen D, Nega B, Solholm A, Farstad M, Bogale N, Graven T, Nielssen NE, Brekke HK, Vikenes K, Haaverstad R. Short-term outcome after open-heart surgery for severe chronic rheumatic heart disease in a low-income country, with comparison with an historical control group: an observational study. Open Heart. 2021 Aug;8(2):e001706. doi: 10.1136/openhrt-2021-001706. PMID 34376574